CLINICAL TRIAL: NCT06353776
Title: MicroPulse Transscleral Laser Therapy and Its Short-term Impact on Ocular Surface
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Walid Zbiba, Professor, University Tunis El Manar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02052023
Record Dates: First submitted 2024-03-25; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Conjunctiva; Cornea
Keywords: MicroPulse; transscleral laser therapy; ocular surface; inflammation; fibrosis; glaucoma
MeSH Terms: conditions — Corneal Diseases; Inflammation; Fibrosis; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MP-TLT + conjunctival biopsy (Experimental): Participants underwent MicroPulse transscleral laser therapy, followed by conjunctival biopsies for the analysis of inflammation and fibrosis.
  Interventions: Procedure: conjunctival biopsy after micropulse transscleral laser therapy

INTERVENTIONS:
Procedure: conjunctival biopsy after micropulse transscleral laser therapy — During MicroPulse TLT, all patients received periocular anesthesia, with an injection of 5 to 10 ml of Lidocaine (Xylocaine 5mg/ml ®) to achieve complete anesthesia.
  The investigators employed the 810 nm Cyclo G6® Laser in its MicroPulse® mode (Iridex Corporation, Mountain View, CA, USA) and delivered laser energy to the eye using the second-generation MicroPulse P3® probe (Iridex Corporation, Mountain View, CA, USA). The laser was calibrated to generate a power output of 2500 mW, and a MicroPulse duty cycle of 31.3%. The curved end of the probe's footplate (bunny ears) was positioned 0.5 to 1 mm away from the corneoscleral limbus, maintaining a perpendicular orientation to the eyeball.
  Following the laser therapy, an immediate conjunctival biopsy measuring 2 * 2 mm and avoiding the laser-treated region was performed.

SUMMARY:
MicroPulse transscleral laser therapy (TLT) is proven to be effective in reducing intraocular pressure with minimal complications in either primary or secondary glaucoma. However, its impact on the human ocular surface remains unexplored. This study aims to bridge this gap by examining the clinical and histopathological effects of MicroPulse TLT on the ocular surface.

DETAILED DESCRIPTION:
This prospective study, conducted at Mohamed Taher Maamouri University Hospital in Nabeul, Tunisia, investigates the clinical and histopathological short-term effects of MicroPulse transscleral laser therapy (TLT) on the ocular surface. The study involves 16 eyes from 15 adult patients. Participants underwent MicroPulse TLT, followed by conjunctival biopsies for the analysis of inflammation and fibrosis. Participants also benefited from ophthalmological examination and responded to the Ocular Surface Disease Index (OSDI) questionnaire before and after MicroPulse TLT.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Non-controlled open-angle glaucoma despite undergoing maximal medical therapy
* Poor therapeutic adherence
* Local or general intolerance to topical treatments.

Exclusion Criteria:

* Ophthalmic or general diseases that could potentially impact the conjunctiva such as symblepharon, ocular injury, or prior eye surgery
* Pevious transscleral laser therapy applied to the same eye
* angle-closure glaucoma
* active ocular inflammation
* a non-functional eye (absence of light perception)
* scleral thinning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
conjunctival inflammation or fibrosis | 1 month
  histological changes of the conjunctiva according to a scale ranging from 0 to 3, with the following interpretation:
  * Grade 0: no difference between the two samples
  * Grade 1: increase in inflammation / fibrosis < 33%
  * Grade 2: increase in inflammation / fibrosis from 33% to 66%
  * Grade 3: increase in inflammation / fibrosis > 66%
intraocular pression | 6 months
  change in intraocular pression
ocular surface disease index score | 6 months
  This score is calculated and ranges from 0 to 100 with the following interpretation:
  * 0 to 12 = Normal
  * 13 to 22 = Mild ocular surface disease
  * 23 to 32 = Moderate ocular surface disease
  * 33 to 100 = Severe ocular surface disease

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Taher Maamouri Hospital, Nabeul, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided